CLINICAL TRIAL: NCT06851598
Title: Safety and Efficacy of Botulinum Toxin-A Injection Into Ischiocavernosus Muscle in Treatment of Premature Ejaculation
Brief Title: Safety and Efficacy of Botulinum Toxin-A Injection Into Ischiocavernosus Muscle for Premature Ejaculation
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abdallah Mohamed Abdallah Mohamed Elgendy (Other)
Responsible Party: Sponsor-Investigator, Abdallah Mohamed Abdallah Mohamed Elgendy, Abdallah Elgendy, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Botox in premature ejaculation
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: 25 units botox
- Group B (Experimental)
  Interventions: Drug: 50 units Botox
- Group C (Experimental)
  Interventions: Drug: 75 units Botox

INTERVENTIONS:
Drug: 25 units botox — 25 units of botox injection into ischiocavernosus muscle
  Arms: Group A
Drug: 50 units Botox — 50 Units botox injection into ischiocavernosus muscle
  Arms: Group B
Drug: 75 units Botox — 75 units botox injection into ischiocavernosus muscle
  Arms: Group C

SUMMARY:
The aim of this work is to assess the efficacy and safety of Botulinum toxin - A injection into ischiocavernosus muscle in treatment of primary premature ejaculation.

DETAILED DESCRIPTION:
Premature ejaculation (PE) is among the most common sexual dysfunctions of men (Porst et al., 2007; Waldinger et al., 2004). It affects more than 50% of men in some populations (Irfan et al., 2020). PE has negative impacts on these men's quality of life, as well as their sexual partners (Rosen & Althof, 2008; Sridharan et al., 2018). The International Society for Sexual Medicine (ISSM) defines PE based on three criteria: the men who have from the first intercourse persistently occurring ejaculation in ≤ 1 min of intercourse (lifelong PE) or significantly reduced ejaculation time (≤ 3 min) later in life (acquired PE), failed to delay ejaculation almost all the time of sexual intercourse, and have developed negative personal and mental conditions (e.g., bother, frustration, distress) and eventually sexual avoidance (Serefoglu et al., 2014). Two types of PE have been widely recognized, ie, lifelong (primary) and acquired (secondary) PE. Lifelong PE is present from the first sexual experience onwards, occurs in almost all attempts at intercourse, and is considered to have a neurobiological etiology. Secondary PE occurs later in life after a period of perceived normal ejaculatory control, and may have a psychological and neurobiological etiology. This type of PE may be triggered by stress or linked to adverse events associated with medications (McCarty E & Dinsmore W, 2012). Treatment of PE varied from behavioral techniques, selective serotonin reuptake inhibitors and local anesthetics with reported variable outcomes, unsatisfactory for many patients (Hanafy S et al.,2019). New lines have been always evolving trying to address this resistant category of patients such as injection of the glans penis with filler (Abdallah H et al.,2012) and neurectomy of the dorsal nerve of the penis (Liu Q et al.,2019). Ejaculation is a spinal cord reflex, which is constituted by emission and expulsion phases (Giuliano F & Clement P,2005). During expulsion, rhythmic contractions of the bulbospongiosus and ischiocavernosus muscles propel semen antegrade through the bulbar and penile urethra. Botulinum-A toxin is a selective blocker of acetylcholine release from nerve endings and inhibits neural transmission when injected into muscle (Whelchel DD et al.,2004). The ischiocavernosus muscle (ICM) encompasses a pair of short pinnate muscles attached to the pelvic ring. This muscle originates at the ischial tuberosity and ends at the crus of the penis while covering the surface of the crus (Hsu GL et al.,2004). The concept of inhibiting stereotyped rhythmic contractions of the bulbospongiosus muscle with Botulinum toxin - A injection for the treatment of lifelong premature ejaculation was initially suggested in 2010 (Serefoglu and Silay, 2010).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with primary (lifelong) PE, with Ejaculation which always or nearly always occurs prior to or within about one minute of vaginal penetration according to The International Society for Sexual Medicine (ISSM) In August 2014.

  _2. Being married for at least 4 months, and in a stable relationship with regular sexual intercourse at least twice per week with a cooperative female partner.
* 3. Normal erectile function.
* 4. Age 18-65 years.

Exclusion Criteria:

1. Erectile dysfunction or other Andrological disorders e.g., Cryptorchidism, Peyronie's disease and 3rd degree varicocele. 2. Major psychiatric or psychological illness. 3. Chronic medical disorders that may limit the usage of Botulinum toxin - A such as myasthenia gravis. 4. Men receiving medications that could affect ejaculatory function e.g., Antidepressants and antihypertensive. 5. Age less than 18 or more than 65.

-

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
IELT(intravaginal ejaculatory latency time) twice weekly | 3 Weeks before and 3 weeks after injection
  With phone stopwatch in seconds twice weekly

CONTACTS AND LOCATIONS:
Overall Officials: Abdelraouf Elmohsen, Professor, Study Chair — Dermatology, Venereology and Andrology Faculty of Medicine, Al-Azhar University; Ahmed Elshahid, Professor, Study Director — Dermatology, Venereology and Andrology Faculty of Medicine, Al-Azhar University
Locations (1):
- Faculty of Medicine, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR